CLINICAL TRIAL: NCT00633516
Title: A Pilot Study to Evaluate the Correlation Between Modified Two Layer Diffuse Optical Spectroscopy With the Clinical and Histological Examinations of Pigmented Skin Lesions Based on Physiological Parameters
Brief Title: A Pilot Study to Evaluate Optical Spectroscopy of Pigmented Skin Lesions
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, David Hsiang, M.D., Division of Surgical Oncology, University of California, Irvine
Other Study IDs: 20086099
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Skin Cancer
Keywords: moles; melanoma
MeSH Terms: conditions — Skin Neoplasms; Nevus; Melanoma | interventions — Spectrum Analysis, Raman

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medical tool: Optical Spectroscopy imaging are Modified Two Layer Diffuse Optical Spectroscopy and multi-spectral imaging and Spatially Modulated Quantitative Spectroscopy
  Interventions: Device: Optical Spectroscopy

INTERVENTIONS:
Device: Optical Spectroscopy — Optical Spectroscopy imaging are Modified Two Layer Diffuse Optical Spectroscopy and multi-spectral imaging and Spatially Modulated Quantitative Spectroscopy
  Other Names: Optical Spectroscopy imaging

SUMMARY:
The incidence of malignant melanoma has increased dramatically in recent decades. In 1930, the lifetime risk of an individual in the United States developing melanoma was 1 in 1,500. This has been exponentially increasing over the years with the risk estimated to be 1 in 75 in 2000 . According to the American Cancer Society, approximately 59,580 new cases of melanoma will be diagnosed in the United States in 2005 and about 7,770 people are expected to die of the disease.

DETAILED DESCRIPTION:
The researcher ucan use special imaging devices to obtain information about a typical mole and melanoma and use this information to determine the different between malignant and benign melanized lesions. The imaging devices are, Modified Two Layer Diffuse Optical Spectroscopy,multi-spectral imaging, and Spatially Modulated Quantitative Spectroscopy can use to measure atypical moles and melanoma and correlate the results of the biopsy tissue histology.

The imaging devices can quantify melanin, oxy and deoxy hemoglobin concentration, water, lipid and reduced scattering coefficients and can compare results to histopathologic. Atypical moles and melanoma have a different optical profile based on physiological parameters compared to benign nevus.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Have atypical mole/s and melanoma

Exclusion Criteria:

* Age less than 18 years old.
* have NO atypical mole/s and melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Measure atypical moles and melanoma | 4 weeks
  Optical Spectroscopy imaging of atypical moles and melanoma to correlate results from the results of the biopsy tissue histology

CONTACTS AND LOCATIONS:
Overall Officials: David JB Hsiang, MD, Principal Investigator — Beckman Laser Institute University of California Irvine; Bruce Tromberg, PhD, Study Director — Beckman Laser Institute University of California Irvine
Locations (2):
- United States (2):
  - Beckman Laser Medical clinic, UCI, Irvine, California
  - UCIMC, Orange, California